CLINICAL TRIAL: NCT06883903
Title: The Effect of Day-Night Cycle on the Transition Time to Full Enteral Feeding in Preterm Newborns Receiving Oropharyngeal Colostrum
Acronym: PRETERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, NEHİR ULU ÖGÜT, NURSE, Biruni University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NEHİR ULU ÖĞÜT
Record Dates: First submitted 2025-02-24; First posted 2025-03-19 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Full Enteral Nutrition; the Day and Night Cycle
Keywords: Preterm; Oropharyngeal Colostrum; Day-Night Cycle; Full Enteral Nutrition; Circadian Rhythm
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: In this study, there are two groups, experimental and control. The experimental group was given a white incubator cover with a white floor, which is routinely used in the daytime unit to create a day/night cycle.
  , dark colored incubator cover was used at night, while the control group received a white incubator with a white floor, which is routinely used in the day/night unit.
  covers were used.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- day-night cycle application (Experimental): In this group, colostrum delivered to the unit within the first 5 days of life was administered by the nurse every three hours for 14 days. In order to create a day/night cycle, a white incubator cover was used routinely in the unit during the day (between 08.00-20.00 hours) and a dark colored incubator cover was used at night (between 20.00-08.00 hours).
  Interventions: Other: day-night cycle application
- routine practice (Active Comparator): In this group, colostrum delivered to the unit within the first 5 days of life was administered every three hours for 14 days by the nurse.
  is the group whose covers are used.
  Interventions: Other: routine practice

INTERVENTIONS:
Other: day-night cycle application — In this group, colostrum delivered to the unit within the first 5 days of life was administered by the nurse every three hours for 14 days. In order to create a day/night cycle, a white incubator cover was used routinely in the unit during the day (between 08.00-20.00 hours) and a dark colored incubator cover was used at night (between 20.00-08.00 hours).
  Arms: day-night cycle application
Other: routine practice — In this group, colostrum delivered to the unit within the first 5 days of life was administered every three hours for 14 days by the nurse.
  is the group whose covers are used.
  Arms: routine practice

SUMMARY:
The aim of this study was to examine the effect of the day-night cycle on the transition time to full enteral nutrition in premature infants receiving oropharyngeal colostrum. The study was conducted with a randomized controlled experimental design to test the potential of an environment that supports the biological rhythms of premature infants to improve feeding processes.

The study was conducted on 60 premature infants born at 28-32 weeks of gestation. Infants were randomly assigned to experimental and control groups, and dark-colored covers were used to create a day-night cycle in the experimental group.

DETAILED DESCRIPTION:
This study was conducted to determine the effect of day-night cycle on the transition of premature newborns receiving oropharyngeal colostrum to full enteral nutrition. The data of the study, which was conducted in a randomized controlled experimental research design between May and December 2022, were collected in the Neonatology Clinic of a university-affiliated training and research hospital in Istanbul after ethical permissions were obtained. The Neonatology Clinic is a level three Neonatal Intensive Care Unit (NICU) and has the capacity to provide specialized care for premature infants.

Sample selection was done using the randomization software at https://www.randomizer.org. As a result of randomization, 30 babies were included in the experimental group and 30 babies were included in the control group. The sample size was calculated using the G*Power 3.1 program, taking into account the findings of similar studies. As a result of this calculation, at least 28 infants were needed for each group and 30 infants were included in both groups, taking into account case losses. Data were obtained from 60 premature newborns who were hospitalized in the Neonatal Intensive Care Unit at 28-32 weeks of gestation and met the inclusion criteria.

The dependent variables of the study were: time to complete enteral nutrition, physiologic parameters (heart rate, oxygen saturation, respiratory rate), discharge time and discharge weight. The independent variable of the study is the day-night cycle established in the Neonatal Intensive Care Unit.

Inclusion Criteria:

Those born between 28-32 weeks of gestation. Infants of parents who agreed to participate in the study. Major congenital anomaly, severe systemic disease, presence of necrotizing enterocolitis, presence of suspected or confirmed sepsis, birth asphyxia (newborns with cord pH/29 arterial pH <7.0).

Newborns admitted to the NICU at ≤ 24 hours of age.

Exclusion Criteria:

Infants excluded from the inclusion criteria for this study Data Collection Forms In the data collection process, Patient Information Form including demographic and clinical information of premature newborns and Patient Monitoring Charts were used to monitor physiologic parameters during the study. In addition, a Voluntary Consent Form was used to obtain written consent from the parents.

Data Collection Tools

The devices used in the study are as follows:

Philips Intellivue MP50 Bedside Monitor: This device was used to measure heart rate, oxygen saturation and respiratory rate of premature infants.

DragerGiraffe Incubator: These are double-walled, digital weighing incubators used to monitor babies in the NICU. These incubators provide a stable environment by preventing the baby from losing heat.

Smart Sensor AS803 DigitalLuxMeter: It was used to measure the light level in the incubator head. Light level control for the babies in the experimental group was provided with this device.

Incubator Covers: Dark colored (navy blue) covers were used in the experimental group to support the day-night cycle. In the control group, standard white covers were used.

Data Collection The families of the premature infants to be included in the study were informed about the purpose, content and method of the study and their written informed consent was obtained. Newborns in both groups were administered 0.1 ml colostrum into the right and left buccal oral cavity at 3-hour intervals for 14 days. In the experimental group, a 12-hour day-night cycle was established with a white incubator cover during the day and a dark colored incubator cover at night. Physiologic parameters of the infants were recorded with monitors before and after the application. In the experimental group, a day-night cycle was achieved by using dark colored covers for the night, while standard white covers were used in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Those born between 28-32 weeks of gestation.
* Infants of parents who agreed to participate in the study.
* Major congenital anomaly, severe systemic disease, necrotizing enterocolitis presence, presence of suspected or confirmed sepsis, birth asphyxia (cord pH / 29 Newborns without arterial pH <7.0).
* Neonates admitted to the NICU at ≤ 24 hours of age.

Exclusion Criteria:

* babies excluded from the inclusion criteria for this study

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Light Meter/Photometer | 14 days, 08.00 am - 20.00 pm
  light source in the neonatal intensive care unit and the area illuminated by the source illumination power analyzes between the Smart Sensor AS803 Digital It is done with Lux Meter device. In the NICU, the lowest light level at the beginning of each incubator 10 lux should be configured with a maximum of 600 lux. The light intensity measured in the incubator in the unit varied between 15 and 40 lx.

SECONDARY OUTCOMES:
Patient Information Questionnaire | baseline
  In the questionnaire prepared to determine the demographic characteristics of premature newborns, questions such as gender, gestational week, mode of delivery, birth weight, hospitalization diagnosis and postnatal age were included. However, it is not a scale.
Patient Follow-up questionnaire | 14 days, 08.00 am - 20.00 pm
  It is a form in which respiratory support status, feeding type, type of food taken, IV fluids given, daily fluid intake/ml, transition to full enteral nutrition are recorded in premature newborns, but it is not a scal

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni Üniversitesi, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Als, H. (2009), Newborn individualized developmental care and assessment program (NIDCAP), New frontier for neonatal and perinatal medicine. J Neonat Perinat Med, 135-47.
- [Background] Altimier., Phillips M.R. (2013), The neonatal ıntegrative developmental care model: seven neuroprotective core measures for family-centered developmental care. Newborn&Infant Nursing Reviews,13, 9-22.
- [Background] Arslan, F., T., Akkoyun, S. (2019), Yenidoğan bütünleştirici gelişimsel bakım modeli: nöroprotektif aile merkezli gelişimsel bakım için yedi temel ölçüm. Ordu Üniversitesi Hemşirelik Çalışmaları, 2(3), 170-1
- [Background] Belfort MB, Anderson PJ, Nowak VA, Lee KJ, Molesworth C, Thompson DK, Doyle LW, Inder TE. Breast Milk Feeding, Brain Development, and Neurocognitive Outcomes: A 7-Year Longitudinal Study in Infants Born at Less Than 30 Weeks' Gestation. J Pediatr. 2016 Oct;177:133-139.e1. doi: 10.1016/j.jpeds.2016.06.045. Epub 2016 Jul 29. PMID 27480198
- [Background] Bilgen, H., S. (2016), Prematürenin enteral beslenmesi. Klinik Tıp Pediatri Dergisi, 8(2), 45-51.
- [Background] Callen J, Pinelli J. A review of the literature examining the benefits and challenges, incidence and duration, and barriers to breastfeeding in preterm infants. Adv Neonatal Care. 2005 Apr;5(2):72-88; quiz 89-92. doi: 10.1016/j.adnc.2004.12.003. PMID 15806448
- [Background] Cohen S, Mandel D, Mimouni FB, Solovkin L, Dollberg S. Gastric residual in growing preterm infants: effect of body position. Am J Perinatol. 2004 Apr;21(3):163-6. doi: 10.1055/s-2004-823778. PMID 15085500
- [Background] Collins CT, Ryan P, Crowther CA, McPhee AJ, Paterson S, Hiller JE. Effect of bottles, cups, and dummies on breast feeding in preterm infants: a randomised controlled trial. BMJ. 2004 Jul 24;329(7459):193-8. doi: 10.1136/bmj.38131.675914.55. Epub 2004 Jun 18. PMID 15208209
- [Background] Damato EG. Research into practice. Measuring stress in pre-term infants. AWHONN Lifelines. 2004 Apr-May;8(2):116-8. doi: 10.1177/1091592304265574. No abstract available. PMID 15137259
- [Background] Efe, Ö., E., Savaşer, S. (2005), Prematüre bebeklerde yalancı emzik uygulamasının total oral beslenmeye geçiş süresine etkisi. Türkiye Klinikleri, (14): 57- 61.
- [Background] Escobar C, Rojas-Granados A, Angeles-Castellanos M. Development of the circadian system and relevance of periodic signals for neonatal development. Handb Clin Neurol. 2021;179:249-258. doi: 10.1016/B978-0-12-819975-6.00015-7. PMID 34225966
- [Background] Esmaeilizadeh, M., Shoja, M., Shoja, E., Shoja, M., Nejat, H., Oudi, D. (2016), Comparing the effects of continuous and cyclical lightings on weight gain and length of hospital stay among preterm neonates. Mod Care J, 13, e8951
- [Background] Fucile S, Gisel E, Lau C. Oral stimulation accelerates the transition from tube to oral feeding in preterm infants. J Pediatr. 2002 Aug;141(2):230-6. doi: 10.1067/mpd.2002.125731. PMID 12183719
- [Background] Greene Z, O'Donnell CP, Walshe M. Oral stimulation for promoting oral feeding in preterm infants. Cochrane Database Syst Rev. 2016 Sep 20;9(9):CD009720. doi: 10.1002/14651858.CD009720.pub2. PMID 27644167
- [Background] Goubet N, Strasbaugh K, Chesney J. Familiarity breeds content? Soothing effect of a familiar odor on full-term newborns. J Dev Behav Pediatr. 2007 Jun;28(3):189-94. doi: 10.1097/dbp.0b013e31802d0b8d. PMID 17565285
- [Background] Grant S, Mayo-Wilson E, Montgomery P, Macdonald G, Michie S, Hopewell S, Moher D; , on behalf of the CONSORT-SPI Group. CONSORT-SPI 2018 Explanation and Elaboration: guidance for reporting social and psychological intervention trials. Trials. 2018 Jul 31;19(1):406. doi: 10.1186/s13063-018-2735-z. PMID 30060763
- [Background] Graven, S., Browne, J, V. (2008), Sensory development in the fetus, neonate, and infant: introductions and overview. Newborn & Infant Nursing Reviews, 8, 169-72.
- [Background] İncekar, Ç., M., Gözen, D. (2019), Preterm bebeklerde bireyselleştirilmiş gelişimsel bakım. Journal of Health and Sport Sciences (JHSS), 2(1), 16-20.
- [Background] Jadcherla SR, Wang M, Vijayapal AS, Leuthner SR. Impact of prematurity and co-morbidities on feeding milestones in neonates: a retrospective study. J Perinatol. 2010 Mar;30(3):201-8. doi: 10.1038/jp.2009.149. Epub 2009 Oct 8. PMID 19812589
- [Background] Johnson AN. Neonatal response to control of noise inside the incubator. Pediatr Nurs. 2001 Nov-Dec;27(6):600-5. PMID 12024534
- [Background] Kenner, C., McGrath, J., M. (2004), Developmental care of newborns and infants. Mosby, Chapter, 14, 260.
- [Background] Küçük, S. (2015), Yenidoğan yoğun bakım ünitelerinde kaliteli uyku. Dokuz Eylül Üniversitesi Hemşirelik Fakültesi Elektronik Dergisi, 8(3), 214-217
- [Background] Laudert S, Liu WF, Blackington S, Perkins B, Martin S, Macmillan-York E, Graven S, Handyside J; NIC/Q 2005 Physical Environment Exploratory Group. Implementing potentially better practices to support the neurodevelopment of infants in the NICU. J Perinatol. 2007 Dec;27 Suppl 2:S75-93. doi: 10.1038/sj.jp.7211843. PMID 18034183
- [Background] Lubbe W. Clinicians guide for cue-based transition to oral feeding in preterm infants: An easy-to-use clinical guide. J Eval Clin Pract. 2018 Feb;24(1):80-88. doi: 10.1111/jep.12721. Epub 2017 Mar 2. PMID 28251754
- [Background] Lucchini R, Bizzarri B, Giampietro S, De Curtis M. Feeding intolerance in preterm infants. How to understand the warning signs. J Matern Fetal Neonatal Med. 2011 Oct;24 Suppl 1:72-4. doi: 10.3109/14767058.2011.607663. Epub 2011 Sep 5. PMID 21892877
- [Background] Long JG, Lucey JF, Philip AG. Noise and hypoxemia in the intensive care nursery. Pediatrics. 1980 Jan;65(1):143-5. No abstract available. PMID 7355011
- [Background] Martin, R., J, Fanaroff, A., A, Walsh, M., C. (2014), Fanaroff and martin's diseases of the fetus and ınfant. Philadelphia: Elsevier Health Science.: NeonatalPerinatal Medicine.
- [Background] McKenna H, Reiss IKM. The case for a chronobiological approach to neonatal care. Early Hum Dev. 2018 Nov;126:1-5. doi: 10.1016/j.earlhumdev.2018.08.012. Epub 2018 Sep 8. PMID 30206009
- [Background] Rodriguez NA, Meier PP, Groer MW, Zeller JM, Engstrom JL, Fogg L. A pilot study to determine the safety and feasibility of oropharyngeal administration of own mother's colostrum to extremely low-birth-weight infants. Adv Neonatal Care. 2010 Aug;10(4):206-12. doi: 10.1097/ANC.0b013e3181e94133. PMID 20697221
- [Background] Parker L, Torrazza RM, Li Y, Talaga E, Shuster J, Neu J. Aspiration and evaluation of gastric residuals in the neonatal intensive care unit: state of the science. J Perinat Neonatal Nurs. 2015 Jan-Mar;29(1):51-9; quiz E2. doi: 10.1097/JPN.0000000000000080. PMID 25633400
- [Background] Pazarcıkcı, F., Efe, E. (2018), Supportive Care Applications From Gavage To Total Oral Feeding In Preterm Infants: Literature Review, 28(3), 92-106.
- [Background] Puntis JW. Nutritional support in the premature newborn. Postgrad Med J. 2006 Mar;82(965):192-8. doi: 10.1136/pgmj.2005.038109. PMID 16517801
- [Background] Sallakh-Niknezhad A, Bashar-Hashemi F, Satarzadeh N, Ghojazadeh M, Sahnazarli G. Early versus Late Trophic Feeding in Very Low Birth Weight Preterm Infants. Iran J Pediatr. 2012 Jun;22(2):171-6. PMID 23056882
- [Background] Shepherd KL, Yiallourou SR, Odoi A, Brew N, Yeomans E, Willis S, Horne RSC, Wong FY. Effects of Prone Sleeping on Cerebral Oxygenation in Preterm Infants. J Pediatr. 2019 Jan;204:103-110.e1. doi: 10.1016/j.jpeds.2018.08.076. Epub 2018 Oct 5. PMID 30297295
- [Background] Tapia-Osorio A, Salgado-Delgado R, Angeles-Castellanos M, Escobar C. Disruption of circadian rhythms due to chronic constant light leads to depressive and anxiety-like behaviors in the rat. Behav Brain Res. 2013 Sep 1;252:1-9. doi: 10.1016/j.bbr.2013.05.028. Epub 2013 May 25. PMID 23714074
- [Background] Vasquez-Ruiz S, Maya-Barrios JA, Torres-Narvaez P, Vega-Martinez BR, Rojas-Granados A, Escobar C, Angeles-Castellanos M. A light/dark cycle in the NICU accelerates body weight gain and shortens time to discharge in preterm infants. Early Hum Dev. 2014 Sep;90(9):535-40. doi: 10.1016/j.earlhumdev.2014.04.015. Epub 2014 May 13. PMID 24831970
- [Background] White-Traut R, Pham T, Rankin K, Norr K, Shapiro N, Yoder J. Exploring factors related to oral feeding progression in premature infants. Adv Neonatal Care. 2013 Aug;13(4):288-94. doi: 10.1097/ANC.0b013e31829d8c5a. PMID 23912022
- [Background] Yiğit, Ş. (2016), Prematüre bebeğin taburcu olduktan sonraki beslenmesi. Klinik Tıp Pediatri Dergisi, 8(2), 52-56.
- [Background] Zee PC, Vitiello MV. Circadian Rhythm Sleep Disorder: Irregular Sleep Wake Rhythm Type. Sleep Med Clin. 2009 Jun 1;4(2):213-218. doi: 10.1016/j.jsmc.2009.01.009. PMID 20160950